CLINICAL TRIAL: NCT02147041
Title: The Effect of Extract of Green Tea on Obese Women Obese Related Hormone Peptides
Brief Title: The Effect of Extract of Green Tea on Obese Women and Obese Related Hormone Peptides
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Chung-Hua Hsu, Chairman of medical affairs, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100XDAA00110; 100XDAA00110 (Other Grant/Funding Number: 100XDAA00110)
Record Dates: First submitted 2014-01-20; First posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus; Hyperlipidemia
Keywords: diabetes mellitus; hyperlipidemia; green tea; epigallocatechin gallate
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias | interventions — Tea; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGCG(Epigallocatechin Gallate) (Experimental): EGCG(Epigallocatechin Gallate)(500 mg, three times a day, 12 weeks)
  Interventions: Drug: EGCG(Epigallocatechin Gallate)
- placebo (Placebo Comparator): cellulose (500mg, three times a day, 12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGCG(Epigallocatechin Gallate) — 500mg, three times a day, duration:12 weeks
  Other Names: EGCG-Epigallocatechin Gallate, green tea extract; cellulose-cellulose
  Arms: EGCG(Epigallocatechin Gallate)
Drug: Placebo
  Arms: placebo

SUMMARY:
The aim of this study is to examine the therapeutic effect of green tea extract on obese women and the correlation analysis between traditional Chinese medicine syndrome and obese related hormone peptides.

DETAILED DESCRIPTION:
Obesity has become a noticeable and worldwide public health problem recently. According to the WHO survey in 2005, 1.6 billion and 400 million adults were found overweight and obese, respectively. In Taiwan, there are more than 30% found overweight in the national survey in 2009. Compare with the ones done in 1999 and 2005, a rising trend of the prevalence of obesity is found. Furthermore, the incidence and prevalence of obesity are also increasing worldwide, especially in the developing and newly industrialized nations. In addition, obesity is related to some chronic diseases, like diabetes mellitus, hyperlipidemia and cardiovascular diseases, which are major lethal health concerns in Taiwan and many developing countries. Taken together, obesity emerges as an important issue lately. The aim of the study is to evaluate the therapeutic effect and safety of green tea extract on demographic characteristics and obesity-related hormone peptide of obese women and to establish an obesity Traditional Chinese Medicine (TCM) syndromes questionnaire, which will undergo well assessing of reliability and validity. Second, we intent to utilize the TCM syndromes and Quality of Life (SF-12, WHO) questionnaire to 200 obesity women for the correlation analysis of TCM syndromes, obesity related hormone peptides and quality of life. The results of this study are expected to assess the effect and safety of green tea extract on obese women and improve the scientific diagnosis of TCM with a quantitative measurement by this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 60 years old women
* Chinese
* body mass index (BMI) > 27 kg/m2
* waist circumference (WC) > 80 cm
* willing to participate in and fill out the questionnaires for this trial.

Exclusion Criteria:

* GPT > 80 U/L, serum creatinine > 2.0 mg/dl
* breast feeding or pregnancy
* heart failure
* acute myocardial infarction
* Stroke
* any other conditions not suitable for trial as evaluated by the physician

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
composite of anthropometric measures | compare between the beginning of the study and after 12 weeks of treatment.
  composite include body weight, waist circumference, hip circumference

SECONDARY OUTCOMES:
Hormone peptide change | compared between the beginning of the study and after 12 weeks of treatment
  hormone peptides such as leptin、adiponectin、ghrelin、fasting insulin resistance、APOB、APOA1
biochemical characteristic change | compare between the beginning of the study and after 12 weeks of treatment.
  blood sugar, creatinine, aminotransferases aspartate, aminotransferases alanine, uric acid and
traditional chinese medicine syndrome classification | compare between the beginning of the study and after 12 weeks of treatment.
  Use questionaire to classify traditional chinese medicine syndrome in obese women
Quality of life evaluation | compare between the beginning of the study and after 12 weeks of treatment.
  (1)12-item Short-Form Health Survey (2)WHOQoL-BREF

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hua Hsu, PHD, Study Chair — Taipei medical hospital, Linsen Chinese Medicine branch
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Result] Hsu CH, Tsai TH, Kao YH, Hwang KC, Tseng TY, Chou P. Effect of green tea extract on obese women: a randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2008 Jun;27(3):363-70. doi: 10.1016/j.clnu.2008.03.007. Epub 2008 May 12. PMID 18468736
- [Derived] Chen IJ, Liu CY, Chiu JP, Hsu CH. Therapeutic effect of high-dose green tea extract on weight reduction: A randomized, double-blind, placebo-controlled clinical trial. Clin Nutr. 2016 Jun;35(3):592-9. doi: 10.1016/j.clnu.2015.05.003. Epub 2015 May 29. PMID 26093535